CLINICAL TRIAL: NCT03024385
Title: Interconception Care at the University of Mississippi Medical Center: An Innovative and Unique Collaborative Continuous Quality Improvement Project Between the Departments of Pediatrics and Family Medicine
Brief Title: Interconception Care at the University of Mississippi Medical Center
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: IMPLICIT Network (Unknown); March of Dimes (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-0116
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Maternal Behavior; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mothers of healthy infants: Mothers of young infants presenting for well child visits between the ages of 0-2 years of age
  Interventions: Behavioral: Well Child Visits

INTERVENTIONS:
Behavioral: Well Child Visits — Mothers of young infants will be screened for maternal behaviors that affect the outcome of future pregnancies. These behaviors are related to the following: family planning; smoking status, prenatal vitamin use and maternal depression. Mothers with positive screens will be offered appropriate resources. This will all take place during the child's routine well-child visit.
  Other Names: Screening questions

SUMMARY:
This model will utilize tools from the IMPLICIT (Interventions to Minimize Preterm and Low Birth Weight Infant through Continuous Quality Improvement Techniques) Network (collaboration of academic family medicine providers). The project involves assessing maternal risk behaviors that significantly affect subsequent birth outcomes: specifically smoking cessation, maternal depression, family planning and preconception folic acid supplementation during well child (WCC) visits. There is evidence that screening mothers for depression can be done at WCC. Data from IMPLCIT network has demonstrated increased screening and referral rates as well as decreased rates of prematurity. This is the first collaborative effort between Pediatrics and Family Medicine.

DETAILED DESCRIPTION:
Specific Aim(s) 1. Determine feasibility of implementing an ICC model as routine standard of care during well child care visits 2. Assess how often physicians routinely implement this model into their practice 3. Increase rates of screening for smoking, depression, folic acid supplementation and family planning during routine visits.

4. Increase rates of referrals for mothers at risk Study Period (inclusive years) This project will take place over a two year period. It will be re-evaluated at monthly intervals to make sure that objectives are being met.

Study Design Study Entry: All mothers presenting with their children to an Ambulatory Pediatric site (North Clinic, Eli Manning and the Pavilion) or Family Medicine (Lakeland and Flowood) for 2 month, 4 month, 6 month, 9 month, 15 month, 18 month and 24 month well child (WCC) visits will be screened for smoking, depression, folic acid supplementation and contraception. Screening will take place at the time of each well child visit. The clinic nurse will present the mother with the screeners for depression and will also ask whether she is smoking, using contraception, and using a folic acid supplementation. Screening scores will be reviewed by the patient's primary care provider. A positive score for PHQ 9 will elicit a referral to Adolescent Medicine and/or Family Medicine for further evaluation. A positive screen for smoking will elicit a referral to the ACT Center at UMMC. Negative responses for contraception use will elicit a referral to Adolescent Medicine and/or Family Medicine for further management. Primary care providers will provide mothers with information and recommendations on folic acid use if they are not using a supplementation.

In Ambulatory Pediatrics mothers in need of services will be referred based on age. Mothers who are 21 years or younger will be referred to Adolescent Medicine. Mothers who are 21 years or older will be referred to Family Medicine. In Family Medicine, mothers will be referred only for depression or smoking cessation.

This project is quality improvement hence screening will be offered to all mothers presenting with their child for well child visits will be screened. Since this project is quality improvement; examining provider behaviors, an exemption from informed consent is requested. Foster parents and non-parental legal guardians will not be screened. Mothers presenting with their child for sick visits will not be screened. Mothers of children older than 2 years of age will not be screened.

All screening will take place at Pediatric primary care sites and at Family Medicine sites, Monday through Friday, from 8am-4pm.

During Phase 2 of the project, mothers of NICU infants will be offered screening. Details of Phase 2 will be presented as an amendment.

Measures: Validated questionnaires will be used to screen depression. Mothers will also be screened regarding smoking, contraceptive use and folic acid supplementation.

Data will be collected monthly as quality improvement reports. Data will be shared with the IMPLICIT Network every 6 months as continuous quality improvement throughout the network.

All de-identified data will be uploaded into REDCap, a password and encrypted database. Data will be shared with March of Dimes to assess progress/process throughout the grant cycle.

On the IMPLICIT REDCap database, site names are listed to facilitate communication and continuous quality improvement monitoring. The IMPLICIT REDCap is maintained on servers at Lancaster General Hospital in Lancaster, Pennsylvania.

Depression Screening: The Patient Health Questionnaire is a validated screening tool for depression. Both forms of the PHQ are graded on a Likert scale, from 0-3 and take just a few minutes to complete. In adults, the PHQ2 has a 97% sensitivity and 67% specificity; the PHQ9 has a 61% sensitivity and 94% specificity. In youth (aged 13-17), the PHQ 9 has 90% sensitivity and 78% specificity. A PHQ9 score of 10 or greater has 88% sensitivity and 88% specificity for major depression. Numeric scoring for PHQ9 is as follows:

Score 5 = Mild Depression Score 10= Moderate Depression Score 15 = Moderately Severe Depression Score 20 = Severe Depression A two item questionnaire (PHQ2) will be given to all mothers of children 2 years or younger presenting for well child visits. If the mother answers yes to either or both of the questions, the screen is scored as positive for depression. The mother will then be screened further with the Patient Health Questionnaire 9 (PHQ9) - a nine item questionnaire.

If the PHQ9 score is positive for moderate depression (10 or greater) the primary care provider will further inquire if the mother is actively suicidal. If so, the primary care provider will send the mother to the Emergency Department for further psychiatric evaluation, as per standard protocol. If the mother is not suicidal, she will be referred to either Adolescent Medicine or Family Medicine Behavioral Health for further evaluation.

Smoking, Contraception and Folic Acid Screening: Screening for smoking, contraception and folic acid supplementation will be "yes or no" items. All scores for mothers will be documented in the child's progress note in the electronic health record.

Inclusion Criteria Mothers who accompany their infants to routine well child care visits will be invited to be screened.

Exclusion Criteria Other legal guardians or foster parents of infants. Mothers of children over 2 years of age will also be excluded.

Number of Subjects (anticipated): This is a feasibility project for quality improvement. It is anticipated that 89 ambulatory care providers will be trained to use this model of ICC. Training will include faculty in general ambulatory pediatrics (8 total) and family medicine (4 total whose practice include pediatric patients). Residents in general pediatrics (47) and family medicine (30) will also be trained.

These providers will have an estimated 1625 unique encounters with mothers. Estimated number of WCC visits for target age group is 13000. Assuming each child gets 8 routine visits in the 1st two years of life (13000/8 =1625).

Outcome Measures Screening and referral rates will be collected and recorded as quality improvement. Current rates of screening and hence referral for these health risks are minimal. It is anticipated that screening rates will initially increase with a subsequent increase in referral rates.

Study Endpoints Current screening and hence referral rates are minimal. This is the first initiative to improve to screening and referral rates. At the end of 2 years, rates of screening for depression, smoking, folic acid supplementation and family planning will be increased to at least 80% of encounter for mothers infants aged 0-2 years of age. Mothers in need of additional intervention will be referred 80% of the time.

Private Health Information Data will be collected in aggregate via chart reviews. Data will be collected by pulling EPIC electronic health record smart-phrases. Private health information will be collected in aggregate. Data pulled from EPIC (infant's name, date of birth, date of visit, ethnicity, medical record number, visit type and demographics) will be de-identified into an internal file and re-coded with a unique REDCap encounter ID. De-identified information will be uploaded into REDCap (a HIPAA secure database) every 6 months. Private health information will not be transmitted to the IMPLCIT REDCap database. REDCap is fully HIPAA compliant.

All 0-2 year well child visits will be pulled and chart review will be done to assess whether screening for depression, contraception, cigarette and folic acid use was performed. Chart review will be performed a monthly basis, at the end of the month. Every 6 months, process of screening will be reviewed and if not at 80% or greater, screening process will be reviewed with all primary care providers.

Data will be assessed for number of positive PHQ9 scores, number of positive smokers and number of mothers not using a contraceptive method or folic acid supplementation.

Data will be assessed for the number of referrals offered to mothers with positive PHQ9 scores, positive smokers and no contraceptive use, to Adolescent Medicine, Family Medicine, Family Medicine Behavioral health or UMMC ACT Center accordingly.

Only de-identified data will be collected (screening rates, questionnaire scores, referral rates). Only the principal investigators and the data analyst (research assistant; a UMMC employee) will have access to the data.

Risks: No identifying information will be collected on any of the screening data to reduce the risk of loss of confidentiality. Mothers are free to withhold any information that they wish to keep confidential.

There are minor risks or discomforts due to participation in this screening. Completion of the screen may be associated with mild distress. Certain screening questions may make participants feel embarrassed or uncomfortable; however, this is a risk that is highly unlikely to be severe given the voluntary participation in the screening.

If such distress occurs for the mother she can discuss with the primary care physician. For mothers who screen positive and are under the age of 18; their guardian will be notified of the recommendation for referral (current standard of care for screening and treatment of minors with depression).

Benefits of Participation in Study:

Subjects: There is a direct benefit to the mother from the screening. Mothers identified as depressed or need of contraceptive services or tobacco cessation will be linked to appropriate services.

Infants/Children: There is an indirect benefit to the children of the mothers screened, such as improved maternal physical and emotional health, which could lead to improved care of the infant/child.

Societal benefits: ICC has been demonstrated to decrease pre-terms births, hence this CQI would ultimately contribute to lower pre-term birth rates in Mississippi

Statistical Methodology Because this is a feasibility study, no formal statistical testing will be performed. Descriptive statistics along with 95% confidence intervals will be used to describe rates of provider screening compliance. In examining the feasibility, we will examine overall rates as well as rates stratified by clinic and age of child.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric Primary Care Providers and Family Medicine Providers at UMMC
2. Mothers of young infants/toddlers who present with their children for well child visits to UMC primary clinics -

Exclusion Criteria:

1. Specialists at UMMC
2. Fathers, grandparents, legal guardians - this screening only applies to mothers of young infants and toddlers -

Ages: 13 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a continuous quality improvement project. It has two aims: can providers screen mothers for health behaviors and can they offer appropriate resources to mothers in need? Thus the study populations are as follows:
  1. Pediatric primary care providers and Family Medicine providers at UMMC
  2. Mothers of young infants/toddlers seen in primary care clinics at UMMC
Sampling Method: Non-Probability Sample
Enrollment: 1625 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Can pediatric primary care provider screen mother for maternal health behaviors during routine well child visits using brief questionnaires? | 2 years
  Pediatric primary care providers (and family medicine providers who care for young infants) will screen mothers for maternal behaviors (smoking status, depression, prenatal multivitamin use, family planning) during routine well child visits of infants aged 0-2 years of age. Mothers will be screened for depression using a validated screening tool (Patient Health Questionnaire or PHQ: the 2 item PHQ-2 will be an initial screen; mothers who have a positive PHQ-2 will be offered the 9-item questionnaire ie the PHQ-9); screening for family planning needs, prenatal multivitamin use and smoking status will be in the form of "yes/no" answers.

SECONDARY OUTCOMES:
Can pediatric primary care providers make appropriate recommendations for mothers with at risk behaviors using brief questionnaires? | 2 years
  Pediatric primary care providers (and family medicine providers who care for young infants) will offer resources for mothers in need of treatment for the following conditions: smoking cessation, depression, multivitamin use, contraception. The Patient Health Questionnaire (PHQ) will be used to screen for depression. The PHQ-2 will be used as an initial screen for depression, mothers who have a positive PHQ-2 will be offered the PHQ-9. Mothers will be screened for suicidal ideation and referred for immediate resources if needed. Mothers who screen positive for depression and not suicidal will be referred to mental health specialists. Mothers will be queried (using "yes/no" responses) with respect to smoking status (mothers will be referred to a smoking cessation program if needed); contraceptive resources will be offered if needed; prenatal vitamins will be recommended if needed. Recommendations will be tracked within the infant's electronic health record.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah MH Jones, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- Univeristy of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MacDorman MF, Mathews TJ. Behind international rankings of infant mortality: how the United States compares with Europe. NCHS Data Brief. 2009 Nov;(23):1-8. PMID 19887034
- [Background] Santos IS, Matijasevich A, Silveira MF, Sclowitz IK, Barros AJ, Victora CG, Barros FC. Associated factors and consequences of late preterm births: results from the 2004 Pelotas birth cohort. Paediatr Perinat Epidemiol. 2008 Jul;22(4):350-9. doi: 10.1111/j.1365-3016.2008.00934.x. PMID 18578748
- [Background] Goedhart G, Snijders AC, Hesselink AE, van Poppel MN, Bonsel GJ, Vrijkotte TG. Maternal depressive symptoms in relation to perinatal mortality and morbidity: results from a large multiethnic cohort study. Psychosom Med. 2010 Oct;72(8):769-76. doi: 10.1097/PSY.0b013e3181ee4a62. Epub 2010 Jul 28. PMID 20668282
- [Background] Johnson K, Posner SF, Biermann J, Cordero JF, Atrash HK, Parker CS, Boulet S, Curtis MG; CDC/ATSDR Preconception Care Work Group; Select Panel on Preconception Care. Recommendations to improve preconception health and health care--United States. A report of the CDC/ATSDR Preconception Care Work Group and the Select Panel on Preconception Care. MMWR Recomm Rep. 2006 Apr 21;55(RR-6):1-23. PMID 16617292
- [Background] Murin S, Rafii R, Bilello K. Smoking and smoking cessation in pregnancy. Clin Chest Med. 2011 Mar;32(1):75-91. doi: 10.1016/j.ccm.2010.11.004. PMID 21277451
- [Background] Sheeder J, Kabir K, Stafford B. Screening for postpartum depression at well-child visits: is once enough during the first 6 months of life? Pediatrics. 2009 Jun;123(6):e982-8. doi: 10.1542/peds.2008-1160. PMID 19482749
- [Background] Ratcliffe S, Gambler A, Gross M, Horst M, Raff T. Preventing Prematurity: One Woman at a Time. The Journal of Lancaster General Hospital. Fall 2012,(7):3;69-74
- [Background] 2015 Premature Birth Report Cards. march of Dimes. http//:www.marchofdimes.org/mission/prematurity-reportcard.aspx. Accessed 2/18/2016
- [Background] Maternal, Infant and Child Health. Healthy People 2020. https://www.healthypeople.gov/2020/topics-objectives/topic/maternal-infant-and-child-health.Accessed 2/18/2016